CLINICAL TRIAL: NCT00746915
Title: A Prospective, Single-Center, Phase I Study Evaluating the Safety and Initial Efficacy of the Epidetect Device for Collection of Bioimpedance Data of Human Tissues in Patients Undergoing Elective Pain Relief Treatment of Lumbar Epidural Steroid Injection Under Fluoroscopy
Brief Title: Phase I Study Evaluating The Safety And Efficacy of a Device for Collection of Electrical Bioimpedance Data
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImpediGuide Ltd (Industry)
Responsible Party: CEO, ImpediGuide Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG-CA001-IS
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: Patients undergoing elective pain relief treatment of lumbar epidural steroid injection under fluoroscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: EpiDetect — During the epidural needle insertion, data will be collected to characterize in real-time the electrical bioimpedance properties of the types of tissue along the path of the needle.

SUMMARY:
The objectives of this study are to evaluate the safety and initial efficacy of the epidural injection procedure when combined with real-time multi-frequency bio-impedance measurements that collect data on the electrical bioimpedance characteristics of living human tissue on the path of the epidural needle.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females 18 - 60 years of age
2. Imaging spine study (CT or MRI) in previous 3 months.
3. American Society of Anesthesiologists (ASA) class I-III
4. Patients undergoing elective standard pain relief treatment of Epidural Steroid Injection
5. Patients must be willing to participate in the study, and provide written informed consent
6. Women of child bearing potential must have a negative pregnancy test during the screening and baseline visits or the patient must be surgically sterile or be at least one year postmenopausal
7. Women of child-bearing potential must be using a medically acceptable method of birth control throughout the study such as: bilateral tubal ligation or the use of either a contraceptive implant, a contraceptive injection, an intrauterine device, or an oral contraceptive that has been taken for at least three months, which the subject agrees to continue using during the study, or a double-barrier method which must consist of a combination of any two of the following: diaphragm, cervical cap, condom or spermicide.

Exclusion Criteria:

1. Any contraindications for epidural injection
2. Patient with severe scoliosis
3. Previous spinal surgery, or any additional surgical intervention in the level of epidural injection other than elective standard pain relief treatment of Epidural Steroid Injection.
4. Documented, known or per examination neurological deficiency in lower extremities.
5. Pregnant or breastfeeding patients
6. Patients who have participated in another study within 30 days of enrolment
7. Investigator's opinion that the patient is medically unfit or would be at major risk if enrolled into the study i.e. known coagulopathy or recent use of anticoagulants or anti aggregates.
8. Presence of fever, sepsis or infection near the point of insertion or an infection in the bloodstream which may "seed" onto the catheter
9. Patients with known Hypovolemia
10. Any known Anatomical abnormalities, such as spina bifida, meningomyelocele or scoliosis
11. Patient suffering problems of the central nervous system, including multiple sclerosis or syringomyelia
12. Patients with identified heart-valve problems
13. Patients excessively hirsute where the surface electrodes are to be placed that are unwilling to shave these areas.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Safety variables collected will include the incidence of adverse events presented by severity, by seriousness and by relationship to study treatment | 2 weeks and 1 month post op

SECONDARY OUTCOMES:
Obtaining real-time bioimpedance measurements in multiple frequencies within the range of 1kHz to 500kHz from human tissues crossed in the epidural needle path. | Day of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Elyad Davidson, Dr., Principal Investigator — Hadassah Medical Oeganization, Ein Kerem
Locations (1):
- Hadassah Medical Organization, Ein Kerem, Jerusalem, Israel